CLINICAL TRIAL: NCT06462820
Title: SAINT® Neuromodulation System for the Treatment of Depression in an Inpatient Setting
Brief Title: SAINT for MDD in an Inpatient Setting Follow-on
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Funding discontinued.
Sponsor: Magnus Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLN-0106
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-10

CONDITIONS: Major Depressive Disorder; Major Depressive Episode; Suicidal Ideation
Keywords: Suicidality; Neuromodulation; Transcranial magnetic stimulation; Depression; Intermittent theta burst stimulation
MeSH Terms: conditions — Depressive Disorder, Major; Suicidal Ideation; Depression

STUDY DESIGN:
Intervention Model Description: Patients will receive either active or sham stimulation to the DLPFC. Patients will be randomized to either condition with a 50:50 chance.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active SAINT Stimulation (Active Comparator): Active SAINT stimulation will be applied to the left dorsolateral prefrontal cortex (DLPFC)
  Interventions: Device: Active SAINT Stimulation
- Sham Stimulation (Sham Comparator): Sham (non-active) stimulation will be applied to the left dorsolateral prefrontal cortex (DLPFC)
  Interventions: Device: Sham SAINT Stimulation

INTERVENTIONS:
Device: Active SAINT Stimulation — Participants who are randomly assigned to this group will receive active SAINT targeted to the left DLPFC. Stimulation intensity will be standardized at 90% of resting motor threshold (adjusted for cortical depth).
  Stimulation will be delivered using the Magventure Magpro X100 TMS system with the Cool-B65 A/P coil.
  Arms: Active SAINT Stimulation
Device: Sham SAINT Stimulation — Participants who are randomly assigned to this group will receive sham stimulation targeted to the left DLPFC.
  Sham stimulation will be delivered using the Magventure Magpro X100 TMS system with the Cool-B65 A/P coil.
  Arms: Sham Stimulation

SUMMARY:
Randomized, multi-site, sham-controlled, double-blinded study

DETAILED DESCRIPTION:
This multi-site, double-blind, randomized, sham-controlled mechanistic trial aims to test the effects of Magnus Neuromodulation System (MNS) with Stanford Accelerated Intermittent Neuromodulation Therapy (SAINT) Technology for the treatment of depression and suicidal cognitions in psychiatrically hospitalized patients with Major Depressive Disorder (MDD) and active suicidal ideation (SI). This will be accomplished by applying the MNS with SAINT protocol (10 applications per day to a customized target within the left dorsolateral prefrontal cortex (L-DLPFC) identified with fMRI for five consecutive days) and measuring changes in depressive symptoms and suicidality at baseline and immediate-post visit.

Th clinical hypothesis is that participants receiving per-protocol active SAINT stimulation will demonstrate a significant difference in Montgomery-Asberg Depression Rating Scale (MADRS) scores/remission rates at the immediate post treatment visit, compared to those who receive per protocol sham SAINT stimulation.

The primary objective of this study is to determine the efficacy of active SAINT vs. sham SAINT in reducing symptoms of depression as measured by the MADRS.

The study will enroll approximately 100 participants and employ a two-arm design with 50 subjects per arm. The target population is adults of all genders and ethnicities who are between 18 and 75 years of age with a diagnosis of treatment-resistant MDD experiencing a current Major Depressive Episode, with active suicidal ideation, and who are otherwise in good general health. Participants must be without contraindications to Magnetic Resonance Imaging (MRI) or transcranial magnetic stimulation (TMS) and must be able to attend all study visits.

This study will deliver both active and sham SAINT via a MagPro X100 edition (MagVenture, Skovlunde, Denmark) TMS device equipped with a Cool-B65 A/P coil. The stimulation paradigm consists of 10 daily sessions (50 total over 5-days) of MNS with SAINT stimulation (3-pulse 50-Hz bursts at 5-Hz for 2-second trains, with trains every 10 seconds), delivered with 50-minute inter-session intervals (10-minute sessions, 50-minutes in between sessions). Stimulation will be delivered at 90% of the resting motor threshold (with depth correction to account for the distance between the scalp and cortex). An operator entered code (derived from the study EDC) will instruct the device to deliver active or sham magnetic stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. Adults of all genders between the ages of 18 and 75 years at the time of screening, who have failed to receive satisfactory improvement from prior antidepressant medication in the current episode
2. Concurrently enrolled in the NIH multi-site trial titled "The Effects of SAINT® Neuromodulation System on Explicit and Implicit Suicidal Cognition"
3. Able to read, understand, and provide written, dated informed consent prior to screening. Proficiency in English sufficient to complete questionnaires/follow instructions during fMRI assessments and SAINT treatments
4. Stated willingness to comply with all study procedures including availability for the duration of the study and to communicate with study personnel about adverse events and other clinically important information
5. Currently diagnosed with Major Depressive Disorder (MDD) and meets criteria for a current Major Depressive Episode (MDE) according to the criteria defined in the Diagnosis and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5)
6. Medical records confirming a history of moderate to severe treatment- resistance as defined by a score of 7-14 on the Maudsley Staging Method153 (MSM)
7. Endorses clinically significant explicit suicidal cognitions (score ≥ 9 on the M-SSI and score ≥ 6 on the BSS self-report)
8. MADRS score of ≥20 at screening (visit 1)
9. rTMS/iTBS naive
10. Access to ongoing psychiatric care before and after completion of the study
11. Access to clinical rTMS after hospital discharge
12. In good general health, as evidenced by medical history
13. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation. Must have a negative urine pregnancy test prior to enrollment

Exclusion Criteria:

1. Pregnancy as confirmed by a positive urine pregnancy test
2. The presence or diagnosis of a prominent anxiety disorder, personality disorder, or dysthymia which in the Investigator's opinion is predominant to MDD
3. Depressed mood/dysphoria as a result of an illness other than MDD (e.g. gender dysphoria)
4. Current severe insomnia (must sleep a minimum of 5 hours each night before stimulation)
5. Current mania or psychosis
6. A history of Bipolar Affective Disorder or Primary Psychotic Disorder
7. Autism Spectrum disorder or Intellectual Disability
8. A diagnosis of obsessive-compulsive disorder (OCD)
9. Current moderate or severe substance use disorder or demonstrating signs of acute substance withdrawal
10. Urine screening test positive for illicit substances
11. Any history of ECT (greater than 8 sessions) without meeting responder criteria
12. Recent (during the current depressive episode) or concurrent use of a rapid acting antidepressant agent (i.e., ketamine or a course of ECT)
13. History of significant neurologic disease, including dementia, Parkinson's or Huntington's disease, brain tumor, unexpected seizure/epilepsy disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma
14. Untreated or insufficiently treated endocrine disorder
15. Contraindications to receiving rTMS (e.g., metal in head, history of seizure, known brain lesion)
16. Contraindications to MRI (ferromagnetic metal in their body)
17. Any current or past history of any physical condition which, in the investigator's opinion, might put the subject at risk or interfere with study results interpretation
18. Treatment with another investigational drug or other intervention within the study period
19. Depth-adjusted SAINT® treatment dose > 65% maximum stimulator output (MSO)
20. Any other condition deemed by the PI to interfere with the study or increase risk to the participant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) Remission Rates | Screening/Baseline, Immediate Post Visit
  Ten item diagnostic questionnaire which psychiatrists use to measure the severity of depressive symptoms in patients with mood disorders.
  We will assess the difference in MADRS scores/remission rates between the per-protocol active SAINT group compared to those who received per-protocol sham treatment at the immediate post treatment visit.

SECONDARY OUTCOMES:
Modified Scale for Suicidal Ideation (M-SSI) | Screening/Baseline, Immediate Post Visit
  A revised version of the Scale for Suicidal Ideation (SSI; Beck et al., 1979). The MSSI is an 18 item scale that contains 13 items from the SSI and 5 additional items.
  We will assess the mean change in the M-SSI from baseline to immediate post treatment visits between the per-protocol active SAINT group compared to those who received per-protocol sham treatment.
Columbia Suicide Severity Rating Scale (C-SSRS) | Screening/Baseline, Immediate Post Visit
  We will use both the Lifetime and the Since Last Visit versions of the C-SSRS to assess suicidality from baseline to immediate post treatment between the per-protocol active SAINT group compared to those who received per-protocol sham treatment.
Montgomery-Asberg Depression Rating Scale (MADRS) Response Rates | Screening/Baseline, Immediate Post Visit
  We will assess the difference in MADRS response rates (reduction >50% of MADRS baseline score) between the per-protocol active SAINT group compared to those who received per-protocol sham treatment at the immediate post treatment visit.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Bentzley, MD, Study Director — Magnus Medical
Locations (4):
- United States (4):
  - University of Iowa, Iowa City, Iowa
  - Weill Cornell Medicine, Manhattan, New York
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas, Ausin - Department of Psychiatry and Behavioral Sciences, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cole EJ, Phillips AL, Bentzley BS, Stimpson KH, Nejad R, Barmak F, Veerapal C, Khan N, Cherian K, Felber E, Brown R, Choi E, King S, Pankow H, Bishop JH, Azeez A, Coetzee J, Rapier R, Odenwald N, Carreon D, Hawkins J, Chang M, Keller J, Raj K, DeBattista C, Jo B, Espil FM, Schatzberg AF, Sudheimer KD, Williams NR. Stanford Neuromodulation Therapy (SNT): A Double-Blind Randomized Controlled Trial. Am J Psychiatry. 2022 Feb;179(2):132-141. doi: 10.1176/appi.ajp.2021.20101429. Epub 2021 Oct 29. PMID 34711062
- [Background] Cole EJ, Stimpson KH, Bentzley BS, Gulser M, Cherian K, Tischler C, Nejad R, Pankow H, Choi E, Aaron H, Espil FM, Pannu J, Xiao X, Duvio D, Solvason HB, Hawkins J, Guerra A, Jo B, Raj KS, Phillips AL, Barmak F, Bishop JH, Coetzee JP, DeBattista C, Keller J, Schatzberg AF, Sudheimer KD, Williams NR. Stanford Accelerated Intelligent Neuromodulation Therapy for Treatment-Resistant Depression. Am J Psychiatry. 2020 Aug 1;177(8):716-726. doi: 10.1176/appi.ajp.2019.19070720. Epub 2020 Apr 7. PMID 32252538
- [Background] Williams NR, Sudheimer KD, Bentzley BS, Pannu J, Stimpson KH, Duvio D, Cherian K, Hawkins J, Scherrer KH, Vyssoki B, DeSouza D, Raj KS, Keller J, Schatzberg AF. High-dose spaced theta-burst TMS as a rapid-acting antidepressant in highly refractory depression. Brain. 2018 Mar 1;141(3):e18. doi: 10.1093/brain/awx379. No abstract available. PMID 29415152